CLINICAL TRIAL: NCT02846142
Title: A Single-center, Randomized, Placebo-Controlled Phase I Study Designed to Assess the Safety, Tolerability, Pharmacokinetics, ECG Effects, Food Effect, and Drug-drug Interaction (DDI) of Hormonal Contraceptives of PTI-428 in Healthy Female Volunteers
Brief Title: Study to Assess the Safety, Tolerability, PK, ECG Effects, Food Effect, and Drug-drug Interaction (DDI) of Hormonal Contraceptives of PTI-428 in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proteostasis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTI-428-02
Record Dates: First submitted 2016-07-18; First posted 2016-07-27 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (7):
- SAD PTI-428 (Active Comparator): The safety, tolerability, and pharmacokinetic profile of PTI-428 will be evaluated following a single dose of PTI-428. Three cohorts are planned for evaluation where subjects will be randomized to PTI-428 or placebo.The subjects will be followed for 7 days post dose.
  Interventions: Drug: PTI-428
- SAD placebo (Placebo Comparator): The safety, tolerability, and pharmacokinetic profile of PTI-428 will be evaluated following a single dose of PTI-428. Three cohorts are planned for evaluation where subjects will be randomized to PTI-428 or placebo.The subjects will be followed for 7 days post dose.
  Interventions: Other: Placebo
- MAD PTI-428 (Active Comparator): Following the conclusion of the respective SAD level dose groups and after sufficient review of study data and approval by the SRC, a second set of healthy adult female subjects will participate in an assigned MAD treatment group. The MAD treatment group is comprised of 3 cohorts. Subjects will be randomized to either PTI-428 or placebo. Each dose will be administered once daily (QD) for a total of 7 days. Follow up visits will occur on Days 12 and 14.
  Interventions: Drug: PTI-428
- MAD placebo (Placebo Comparator): Following the conclusion of the respective SAD level dose groups and after sufficient review of study data and approval by the SRC, a second set of healthy adult female subjects will participate in an assigned MAD treatment group. The MAD treatment group is comprised of 3 cohorts. Subjects will be randomized to either PTI-428 or placebo. Each dose will be administered once daily (QD) for a total of 7 days. Follow up visits will occur on Days 12 and 14.
  Interventions: Other: Placebo
- OC (ethinyl estradiol and levonorgestrel) DDI Period A (Experimental): Treatment period A will consist of once daily oral contraceptive (OC) for 28-days (21-day hormonal active + 7 days off).
  Interventions: Drug: ethinyl estradiol and levonorgestrel
- OC (ethinyl estradiol and levonorgestrel) DDI Period B (Active Comparator): Treatment period B will randomize subjects to PTI-428 or placebo in combination with once daily OC daily for 28 days (21-day hormonal active + 7 days off).
  Interventions: Drug: PTI-428; Drug: ethinyl estradiol and levonorgestrel
- OC (ethinyl estradiol and levonorgestrel) DDI (Placebo Comparator): Treatment period B will randomize subjects 4:1 to PTI-428 or placebo in combination with once daily OC daily for 28 days (21-day hormonal active + 7 days off).
  Interventions: Other: Placebo; Drug: ethinyl estradiol and levonorgestrel

INTERVENTIONS:
Drug: PTI-428
  Arms: MAD PTI-428; OC (ethinyl estradiol and levonorgestrel) DDI Period B; SAD PTI-428
Other: Placebo
  Arms: MAD placebo; OC (ethinyl estradiol and levonorgestrel) DDI; SAD placebo
Drug: ethinyl estradiol and levonorgestrel
  Arms: OC (ethinyl estradiol and levonorgestrel) DDI; OC (ethinyl estradiol and levonorgestrel) DDI Period A; OC (ethinyl estradiol and levonorgestrel) DDI Period B

SUMMARY:
This trial will consist of three parts: the first two parts will enroll healthy female volunteers into a single ascending dose (SAD) and multiple ascending dose (MAD) treatment groups.

The SAD treatment group is comprised of at least 3 cohorts where subjects will be randomized to a single dose of either PTI-428 or placebo and will be followed for 7 days post dose. A total of 24 subjects are anticipated to participate in this part of the study.

Following the conclusion of the respective SAD level dose groups and after sufficient review of study data and approval by the SRC, a second set of healthy adult female subjects will participate in an assigned MAD treatment group. The MAD treatment group is comprised of 3 cohorts where subjects will be randomized to either PTI-428 or placebo and will be followed for a total of 14 days. The SRC will convene after the completion of each cohort to evaluate safety, PK and other relevant data. The SRC will determine whether to proceed to the next planned dose level, to reduce the dose, or to stop the study. The next cohort may commence only after written SRC approval. A total of 24 subjects are anticipated to participate in this part of the study.

Following completion of the SAD and MAD, 40 female healthy volunteers will participate in two treatment periods of the DDI study component: Treatment period A will consist of once daily oral contraceptive (OC) for 28-days (21-day hormonal active + 7 days off).

Treatment period B will randomize subjects to PTI-428 or placebo in combination with once daily OC for 28 days (21-day hormonal active and PTI-428 or placebo + 7 days off). Following completion of the subjects' second treatment period, they will be followed for 7-days after their last dose.

ELIGIBILITY:
Inclusion Criteria:

* Adult females age 18 - 55 years old, inclusive, at the time of informed consent.
* For the DDI Oral Contraceptive Cohort, women of child bearing potential with intact ovarian function by medical history and history of regular menstrual. cycles.
* Body mass index (BMI) ≥18 < 30 kg/m2.
* Subject must be non-smoker and non-tobacco user for a minimum of 30 days prior to screening and for the duration of the study.
* Subject understands the full nature and purpose of the study, including possible risks and side effects, and is willing and able to comply with all compulsory study procedures and provides informed consent/permission prior to any study procedures being performed.

Exclusion Criteria:

* History or current evidence of any clinically significant cardiac, endocrinologic, hematologic, hepatobiliary, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the Investigator.
* Abnormal liver function as defined by:
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) or bilirubin > 1.5 x upper limit of the normal range.
* Abnormal renal function at screening defined as:
* Creatinine clearance < 80mL/min using the Cockroft-Gault equation.
* No clinically significant screening results that would exclude subject from the study (e.g., medical histories, physical examination, ECGs, vital signs,and laboratory profiles) as deemed by the investigator.
* Platelet count < 150,000 cell/mm3
* Participation in another clinical trial or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer, prior to Study Day 1.
* History of cancer within the past five years (excluding non-melanoma skin cancer).
* History of alcohol or drug abuse or dependence within 12 months of screening as determined by the Investigator.
* Positive urine screen for prohibited drugs (cocaine, cannabinoids, nicotine [urine cotinine is the detection mechanism for nicotine], opiates, barbiturates, amphetamines, and benzodiazepines) or positive alcohol test at screening.
* Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (HCVAb).
* Clinically significant infection within 3 months of screening as determined by the Investigator.
* Known or suspected hypersensitivity or idiosyncratic reaction to study medication or any components thereof.
* Has donated blood within 3 months of screening or plans to donate blood within 3 months of study completion.
* Pregnant or nursing women.
* Any conditions that, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study.
* Females of child-bearing potential, unless they are willing to use highly effective methods of contraception during participation in the clinical study and for 30 days after termination from study.
* Use of prohibited medications within 14 days prior to dosing of study drug.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
SAD and MAD: Safety and tolerability measured by number of subjects who experience adverse events and potential clinically significant changes in safety labs, electrocardiograms (ECGs), physical examinations, and vital signs | baseline to 7 days
SAD: Apparent terminal half-life (t1/2) of single oral dose | through 72-hours post dose
SAD: Time to reach maximum plasma concentration (Tmax) of single oral dose | through 72-hours post dose
SAD: Maximum plasma concentration (Cmax) of single oral dose | through 72-hours post dose
SAD: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUC0-t) of single oral dose | through 72-hours post dose
MAD: Apparent terminal half-life (t1/2) of multiple oral doses | through 72 hours post day 7 dose
MAD: Time to reach maximum plasma concentration (Tmax) of multiple oral doses | through 72 hours post day 7 dose
MAD: Maximum plasma concentration (Cmax) of multiple oral doses | through 72 hours post day 7 dose
MAD: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUC0-t) of multiple oral doses | through 72 hours post day 7 dose
SAD: Cumulative amount of PTI-428 excreted unchanged in urine (Ae) | through 72-hours post dose
SAD: renal clearance (CLR) | through 72-hours post dose
MAD: Cumulative amount of PTI-428 excreted unchanged in urine (Ae) | through 72 hours post day 7 dose
MAD: renal clearance (CLR) | through 72 hours post day 7 dose
OC: Time to reach maximum plasma concentration (Tmax) of multiple oral doses | through day 49
OC: Maximum plasma concentration (Cmax) of multiple oral doses | through day 49
OC: Area under the concentration-time curve from time 0 to time of last measurable concentration (AUC0-t) of multiple oral doses | through day 49

CONTACTS AND LOCATIONS:
Locations (1):
- Overland Park, Kansas, United States